CLINICAL TRIAL: NCT03690544
Title: A Pilot Study Evaluating the Efficacy of Apremilast in the Treatment of Subjects With Severe Recurrent Aphthous Stomatitis (RAS)
Brief Title: Apremilast for RAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Alison J. Bruce, Principle Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-002914
Record Dates: First submitted 2018-09-04; First posted 2018-10-01 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Aphthous Stomatitis
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: Apremilast 30mg orally twice daily for 16 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Apremilast 30mg orally twice daily for 16 weeks, sixteen weeks on active study. Post treatment follow-up period of 8 weeks, in the Treatment of Subjects with Severe Recurrent Aphthous Stomatitis (RAS)
  Interventions: Drug: Apremilast 30mg

INTERVENTIONS:
Drug: Apremilast 30mg — Apremilast is an oral small-molecule inhibitor of phosphodiesterase (PDE) 4 that works intracellularly to modulate a network of pro-inflammatory and anti-inflammatory mediators. PDE 4 is a cyclic adenosine monophosphate (cAMP)-specific PDE and the dominant PDE in inflammatory cells. PDE4 inhibition elevates intracellular cAMP levels, which in turn down-regulates the inflammatory response by modulating the expression of TNF-alfa, IL-23, IL-17 and other inflammatory cytokines. Cyclic AMP also modulates levels of anti-inflammatory cytokines such as IL-10. Apremilast has immunomodulatory activity and, therefore, has the potential to be effective in the treatment of RAS.

SUMMARY:
Determination of treatment efficacy and safety of Apremilast in patients with RAS

DETAILED DESCRIPTION:
The study will be a pilot study using apremilast 30mg orally twice daily, for treatment of RAS in males and females between 18 and 70 years old.

Subjects will be recruited from the clinical practice of the Department of Dermatology or Division of Rheumatology at Mayo Clinic Florida. Fifteen males and females with RAS will be enrolled.

The study will consist of 3 phases: a screening phase, a 16 week treatment phase and an 8 week posttreatment observational follow-up phase.

The screening phase will consist of: obtaining informed consent, demographic information, medical history, inclusion and exclusion criteria, prior and concomitant medication use, adverse events; collecting vital signs and weight; performing complete physical examination and limited physical examination; obtaining hematology, serum chemistry, urinalysis, pregnancy test and providing contraception education.

During the 16-week treatment phase, all subjects receive apremilast.

All subjects who complete the active treatment phase are to enter the 8-week posttreatment observational follow-up phase.

ELIGIBILITY:
Inclusion Criteria

1. Male and female subjects between 18 and 70 years of age
2. Oral ulcers that occurred at least monthly in the 6 month period prior to enrollment
3. Had at least 2 oral ulcers in the 4 weeks prior to enrollment at baseline
4. At least 3 oral ulcers during an ulcer flare
5. Patients must be candidates for systemic therapy for the treatment of oral ulcers, those that are considered unsuitable for topical therapy alone based on severity of disease, or whose oral ulcers cannot be adequately controlled with topical therapy.
6. Female premenopausal subjects must use one of the approved contraceptive options while taking apremilast and for at least 28 days after administration of the last dose of apremilast
7. Patients are able and willing to provide written informed consent after the nature of the study is fully explained.
8. No evidence of systemic disease

Exclusion Criteria

1. Prior use of apremilast.
2. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
3. Having received concomitant immune modulating therapy 12 weeks prior to enrollment, systemic steroids 6 weeks prior to enrollment or topical steroids within 4 weeks prior to enrollment.
4. Pregnant women or breast-feeding mothers.
5. Systemic or opportunistic fungal infection.
6. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (tuberculosis and atypical mycobacterial disease, hepatitis B and C and herpes zoster, histoplasmosis, coccidiomycosis) or any major episode of infection requiring hospitalization or treatment with IV or oral antibiotics within 4 weeks of the screening phase.
7. History of positive test for, or any clinical suspicion of, human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency.
8. History of depression.
9. Malignancy or history of malignancy, except for:

   a - treated (ie, cured) basal cell or squamous cell in situ skin carcinomas; b - treated (ie, cured) cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
10. Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
11. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
12. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
13. Active substance abuse or a history of substance abuse within 6 months prior to screening.
14. Presence of any of the following vitamin deficiencies - B1, B2, B6, B12, vitamin C, zinc, folate, iron.
15. Celiac disease.
16. Inflammatory Bowel Disease.
17. Genital aphthous ulcers.
18. Behçet's disease.
19. History of positive patch test for allergic contact stomatitis.
20. Positive anti-endomysial or anti-gliadin antibodies.
21. A diagnosis of uveitis (current or previous).
22. Erythema nodosum-like lesions (current or previous).
23. An established diagnosis of a systemic disease (SLE, Reiter's, Sweet's and MAGIC syndrome).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Bruce, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Subjects received Apremilast 30mg orally twice daily for 16 weeks, sixteen weeks on active study. Post treatment follow-up period of 8 weeks, in the Treatment of Subjects with Severe Recurrent Aphthous Stomatitis (RAS)
  Apremilast 30mg: Apremilast is an oral small-molecule inhibitor of phosphodiesterase (PDE) 4 that works intracellularly to modulate a network of pro-inflammatory and anti-inflammatory mediators. PDE 4 is a cyclic adenosine monophosphate (cAMP)-specific PDE and the dominant PDE in inflammatory cells. PDE4 inhibition elevates intracellular cAMP levels, which in turn down-regulates the inflammatory response by modulating the expression of TNF-alfa, IL-23, IL-17 and other inflammatory cytokines. Cyclic AMP also modulates levels of anti-inflammatory cytokines such as IL-10. Apremilast has immunomodulatory activity and, therefore, has the potential to be effective in the treatment of RAS.
Period: Overall Study
Arm/Group | Single Arm
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 56 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  Hispanic or Latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Duration of RAS Lesions
Description: The total length of time (duration) subjects experienced RAS lesions. Measured in weeks
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Single Arm
Number analyzed (Participants) | 15
weeks | 1.57 (0.68)

2. Primary Outcome: Change in Number of RAS Lesions
Description: Number of participants with fewer oral ulcers at Week 24 compared to Baseline
Time Frame: baseline, 24 weeks
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 15
participants | 11

3. Primary Outcome: Duration of the Remission Period Between Ulcer Episodes
Description: The length of time of remission of RAS lesions experienced by the subjects. As measured in months.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Single Arm
Number analyzed (Participants) | 15
months | 2.00 (0.85)

4. Secondary Outcome: Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 15
Participants | 11

5. Secondary Outcome: Discontinuation of Study Participants
Description: Number of subjects who prematurely discontinue treatment with apremilast due to any adverse event.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 15
Participants | 3

6. Secondary Outcome: Change in Visual Analog Scale Pain Score (VAS) From Baseline to 16 Weeks and Baseline to 24 Weeks.
Description: The Visual Analog Scale (VAS) for Pain is a validated tool used to measure pain. A 100mm horizontal line anchored by "no pain" (score of 0) and "pain as bad as it could be" (score of 100).
Time Frame: baseline, 16 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 15
units on a scale
  baseline to 16 weeks | -4 (3.0)
  baseline to 24 weeks | -2 (4.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately 24 weeks
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=15)
Nausea (General disorders) | 9
Diarrhea (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03690544/Prot_SAP_000.pdf